CLINICAL TRIAL: NCT01794013
Title: A Randomized Controlled Trial of DIR/ Floortime™ Parent Training Intervention for the Children With Developmental Disabilities
Brief Title: DIR/ Floortime™ Parent Training Intervention for the Children With Developmental Disabilities
Acronym: RCT/DD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kingkaew Pajareya (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor-Investigator, Kingkaew Pajareya, Faculty of Medicine Siriraj Hospital, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si089/2013
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Cerebral Palsy; Down's Syndrome; Delayed Development
Keywords: Parent training; DIR/ Floortime Approach; Children with developmental disabilities
MeSH Terms: conditions — Cerebral Palsy; Down Syndrome; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent trianing (Active Comparator): The parent training group will learn about DIR/ Floortime™ model approach through one on one coaching for 1 hour at the beginning of the study, the end of 1st and 3th month and through 2 hours DVD lecture and a pocket book.
  Interventions: Behavioral: Parent training
- Routine care (Active Comparator): The children in the control group will continue their standard routine care.
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Parent training — All parents in the intervention group had to learn about DIR/ Floortime™ model approach through one on one coaching (1 hour/ session for three sessions) and through 2 hours DVD lecture.
  Other Names: DIR/ Floortime parent training
  Arms: Parent trianing
Behavioral: Routine care — routine care
  Arms: Routine care

SUMMARY:
The objective of this study is to test whether adding the parent training program using the relationship-based approach could help the children with development disabilities (DDs) would confer additional benefits over routine clinical care available to both groups in terms of improving their development and reducing behavior problems.

DETAILED DESCRIPTION:
The objective of this study is to test whether adding the parent training program using the relationship-based approach could help the children with development disabilities (DDs) would confer additional benefits over routine clinical care available to both groups in terms of improving their development and reducing behavior problems.

The study treatment involves intervention entirely with parents of children with DDs, rather than directly with the children themselves. Before the first session, all parents in the intervention group had to learn about DIR/ Floortime™ model approach through 1 - hour one on one coaching (at the beginning oft the study, the end of 1st and 3rd month) and through 2 hours DVD lecture and a pocket book. The parent in the intervention group will be asked to carry out FloortimeTM together with using Floortime strategies during daily activities a minimum of 15 hour per week. Meanwhile, the children in the control groups will continue their routine care. The baseline assessment and follow up time schedule were similar to those of the intervention group.

ELIGIBILITY:
Inclusion Criteria:

The children with developmental disabilities :

1. age between 2 - 6 years of age
2. ambulatory
3. living with the primary caregiver for at least 6 months.

Exclusion Criteria:

The children are excluded if :

1. autism
2. deaf
3. blind
4. serious medical problems (e.g. severe congenital heart disease, intractable seizure (a seizure frequency of at least one attack per month during six months despite receiving two anticonvulsant drugs)
5. their parents : not literate, has known chronic psychiatric, or physical illness

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The change in The Child Behavior Rating Scale (CBRS) | 4 months

SECONDARY OUTCOMES:
The change in The Functional Emotional Developmental Questionnaire (FEDQ) | 4 months

OTHER OUTCOMES:
The change in The Mullen Scales of Early Learning (MSEL) | 4 months
The change in The Parenting Stress Index-Short Form (PSI-SF) | 4 months
Client's Satisfaction | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kingkaew Pajareya, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Kingkaew Pajareya, Bangkok, Thailand